CLINICAL TRIAL: NCT02658045
Title: A Clinical Evaluation of the Oxitone Non-invasive Oximeter. Method Comparison Study vs. a Standard Clinical Pulse-oximeter Monitor. A Prospective Open Study
Brief Title: A Clinical Evaluation of the Oxitone Non-invasive Oximeter
Acronym: CPOM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0172-15MMC
Record Dates: First submitted 2015-12-02; First posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-11

CONDITIONS: COPD; Chronic Lung Disease
Keywords: oxygen saturation; monitoring; oximeter
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal healthy volunteers: Measurement of oxygen saturation simultaneously by standard oximeter and Oxitone oximeter in healthy volunteers during 6 min walking test
  Interventions: Device: Standard Oximeter; Device: Oxitone oximeter
- COPD patients: Measurement of oxygen saturation simultaneously by standard oximeter and Oxitone oximeter in COPD patients during 6 min walking test
  Interventions: Device: Standard Oximeter; Device: Oxitone oximeter

INTERVENTIONS:
Device: Standard Oximeter — Oxygen saturation will be measured by standard oximeter
Device: Oxitone oximeter — Oxygen saturation will be measured by Oxitone oximeter

SUMMARY:
The trial shall assess the accuracy of the Oxitone® 1000 in measuring oxygen saturation, by comparing its measurement to reference devices: non-invasive SpO2 and pulse-rate values determined by a pulse oximeter. A total of approximately 40 subjects: 20 healthy and 20 COPD (chronic obstructive pulmonary disease ) patients will be enrolled. These subjects will be enrolled at the medical center pulmonary department and will be recruited from the clinic patient base. The subjects will be represented by male and female adults who optimally cover a range of ethnic backgrounds (skin pigmentation). All testing will be performed in singleton and in a blinded fashion. This study will be conducted with the approval of the medical center ethics committee.

This is a comparison open study with no subject follow-up.

DETAILED DESCRIPTION:
The Oxitone® 1000 oximetry readings are accurate and measure with an acceptable relative absolute difference (RAD) when compared to accepted measurement systems (FDA recognized predicate) the "Reference".

The objectives:

1. To validate the Oxitone® 1000 performance in continuous or spot oximetry monitoring, relative to Reference readings.
2. To aggregate longitudinal clinical data from COPD patients measuring SpO2, pulse rate and activity.
3. To evaluate the main device parameters and characteristics such as sensor placement tolerance, device accuracy, precision, convenience and easy-to-use at stationary supine or seated tests and at mild motions as well.
4. To determine whether the measured data provided from patients (SpO2, pulse rate and movement) is useful in adjusting their treatment protocol.
5. To assess the safety and tolerability (compliance) of the Oxitone® 1000 in continuous oximetry monitoring in order to obtain sufficient clinical trial data in order to define performance criteria of the device system that are acceptable / useful in the medical context for patient populations and other healthy individuals, in which the device is likely to be used.

Overview: The trial shall assess the accuracy of the Oxitone® 1000 in measuring oxygen saturation, by comparing its measurement to reference devices: non-invasive SpO2 and pulse-rate values determined by a pulse oximeter. A total of approximately 40 subjects (20 healthy and 20 COPD patients) will be enrolled. These subjects will be enrolled at the medical center pulmonary department and will be recruited from the clinic patient base. The subjects will be represented by male and female adults who optimally cover a range of ethnic backgrounds (skin pigmentation). All testing will be performed in singleton and in a blinded fashion. This study will be conducted with the approval of the medical center ethics committee.This is a comparison open study with no subject follow-up.

Procedure: All instruments will be checked for functionality and battery operational capacity, prior to subject attachment including the data collection system, i.e. the wireless (B.T.) connectivity to P.C. (synchronized bidirectional two channels).

The "Reference" oximeter device shall be set for averaging mode of 12 seconds. Two sensors will be placed simultaneously on the subjects: A standard SpO2 (reference) will be placed on the subject's index finger and the tested Oxitone® 1000 will be placed on the subject's wrist of the same hand.

Methods:: The investigators are to study approximately 40 subjects, both normal, i.e. comparison group and patients with a variety of pulmonary conditions that effect oxygen saturation. The investigators will compare the oxygen saturation of each subject as measured with Oxitone® 1000 device and with the oxygen saturation as measured with calibrated conventional FDA approved pulse oximeter (predicate). The "Reference". No treatment decision will be made utilizing the results of the tested device.

Trial design:

A. Healthy subjects: Spot-check measurements of 20 healthy volunteers simultaneously tested by using Oxitone oximeter and standard fingertip pulse oximeter at stationary state i.e. at sitting and standing positions up to 6 minutes each.

1. A 6-minute.walk: oximetry tests of 20 healthy volunteers simultaneously tested using Oxitone oximeter and standard fingertip pulse oximeter in accordance with the industry (Medical) standards of 6-min walk protocol. Measurements are collected and recorded continuously prior to test, during the test and after 6 minutes the test. The distance of the 6-min walk will be recorded (CRF).

B. COPD (Chronic obstructive pulmonary disease) subjects

1. Spot-check measurements up to 20 ambulatory COPD patients. Patients should be referred and admitted to the pulmonary lab for clinical treatment or should be under the rehabilitation procedures. Measurements will be made simultaneously using Oxitone® oximeter and while standard fingertip pulse oximeter stationary state at e.g. supine or dorsal elevated sitting, and while standing (upright) positions up to 6 min each.
2. A 6-min walk oximetry tests of ambulatory COPD patients. Patients should be referred to the pulmonary lab for clinical purposes or should be under the rehabilitation procedures. The measurements are taken using Oxitone® oximeter and standard fingertip pulse oximeter in accordance with the standard protocol. Measurements are taken continuously prior to the test, during the test and 1 minute after the test, at rest. The distance of the 6-min walk will be recorded. Rehabilitation subjects procedures. The measurements are taken using Oxitone® Oximeter and standard fingertip pulse oximeter in accordance with the standard protocol. Measurements are taken continuously prior to the test. The distance of the 6-min walk will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary sick and healthy male and female volunteers aged 18 years and over (any race or ethnicity).
* Subjects who are willing to give informed consent.
* No precautions are required: this study involves no known additional risk to the subjects.

Exclusion Criteria:

* Participants under the age of 18 years
* Significant deformity, degenerative changes or edema of the hand wrist
* Localized infection, ulceration or skin breaks involving the wrist
* Vascular disease or Raynaud's phenomenon affecting the hand
* Participants who are unable to give informed written consent
* Anemia: Hb < 10.0 g/dl

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 30 subjects will be recruited. Participants will be screened for inclusion/exclusion criteria at enrolment and will be asked to sign an informed consent form. Only those who give written informed consent will be included in the study. Basic clinical, demographic including skin type (Fitzpatrick scale) information and past medical history (CRF) will be recorded.
  Patient selection: Adult patients over the age of 18 of both genders will be recruited. Patients will be either outpatients in the pulmonary department, or ambulatory patients undergoing rehabilitation.
  Normal Healthy volunteers will be recruited from hospital personnel or medical students. There will be no known additional risk for the subjects.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
change in oxygen saturation from baseline to six minute walk | Baseline and after six minute walk
  Oxygen saturation is measured with standard oximeter and Oxitone oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Alex 1 Guber, MD, Principal Investigator — Meir Medical Center

REFERENCES:
- [Background] Hornberger C, Matz H, Konecny E, Frankenberger H, Bonk R, Avgerinos J, Benekos K, Valais J, Ikiades A, Gil-Rodriguez J, Wouters P, Meyfroidt G, Ponz L, Gehring H. Design and validation of a pulse oximeter calibrator. Anesth Analg. 2002 Jan;94(1 Suppl):S8-12. PMID 11900044
- [Background] Mendelson Y. Pulse oximetry: theory and applications for noninvasive monitoring. Clin Chem. 1992 Sep;38(9):1601-7. PMID 1525987
- [Background] Trivedi NS, Ghouri AF, Shah NK, Lai E, Barker SJ. Effects of motion, ambient light, and hypoperfusion on pulse oximeter function. J Clin Anesth. 1997 May;9(3):179-83. doi: 10.1016/s0952-8180(97)00039-1. PMID 9172022